CLINICAL TRIAL: NCT05174637
Title: A PhaseⅠStudy to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of FDA018-ADC in Patients With Advanced Solid Tumors
Brief Title: A Study of FDA018-ADC in Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: F0024-101
Record Dates: First submitted 2021-11-16; First posted 2022-01-03 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Advanced/ Metastatic Solid Tumors
Keywords: Trop-2; Solid tumor; TNBC; Antibody-drug conjugate, ADC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- FDA018-ADC A mg/kg (Experimental): Subjects will receive FDA018-ADC A mg/kg of body weight via intravenous (IV) infusion on Day 1 of a 14-Day cycle (Cycle 1) and on Day 1 and 8 of a 21-day cycle (Cycle 2 ~ Cycle n) in dose escalation phase, and on Day 1 and 8 of a 21-day cycle(Cycle 1 ~ Cycle n) in dose expansion phase, until the date of first documented progression or unacceptable toxicity or death.
  Interventions: Drug: FDA018-ADC
- FDA018-ADC B mg/kg (Experimental): Subjects will receive FDA018-ADC B mg/kg of body weight via intravenous (IV) infusion on Day 1 of a 14-Day cycle (Cycle 1) and on Day 1 and 8 of a 21-day cycle (Cycle 2 ~ Cycle n) in dose escalation phase, and on Day 1 and 8 of a 21-day cycle(Cycle 1 ~ Cycle n) in dose expansion phase, until the date of first documented progression or unacceptable toxicity or death.
  Interventions: Drug: FDA018-ADC
- FDA018-ADC C mg/kg (Experimental): Subjects will receive FDA018-ADC C mg/kg of body weight via intravenous (IV) infusion on Day 1 of a 14-Day cycle (Cycle 1) and on Day 1 and 8 of a 21-day cycle (Cycle 2 ~ Cycle n) in dose escalation phase, and on Day 1 and 8 of a 21-day cycle(Cycle 1 ~ Cycle n) in dose expansion phase, until the date of first documented progression or unacceptable toxicity or death.
  Interventions: Drug: FDA018-ADC
- FDA018-ADC D mg/kg (Experimental): Subjects will receive FDA018-ADC D mg/kg of body weight via intravenous (IV) infusion on Day 1 of a 14-Day cycle (Cycle 1) and on Day 1 and 8 of a 21-day cycle (Cycle 2 ~ Cycle n) in dose escalation phase, and on Day 1 and 8 of a 21-day cycle(Cycle 1 ~ Cycle n) in dose expansion phase, until the date of first documented progression or unacceptable toxicity or death.
  Interventions: Drug: FDA018-ADC
- FDA018-ADC E mg/kg (Experimental): Subjects will receive FDA018-ADC E mg/kg of body weight via intravenous (IV) infusion on Day 1 of a 14-Day cycle (Cycle 1) and on Day 1 and 8 of a 21-day cycle (Cycle 2 ~ Cycle n) in dose escalation phase, and on Day 1 and 8 of a 21-day cycle(Cycle 1 ~ Cycle n) in dose expansion phase, until the date of first documented progression or unacceptable toxicity or death.
  Interventions: Drug: FDA018-ADC
- FDA018-ADC F mg/kg (Experimental): Subjects will receive FDA018-ADC F mg/kg of body weight via intravenous (IV) infusion on Day 1 of a 14-Day cycle (Cycle 1) and on Day 1 and 8 of a 21-day cycle (Cycle 2 ~ Cycle n) in dose escalation phase, and on Day 1 and 8 of a 21-day cycle(Cycle 1 ~ Cycle n) in dose expansion phase, until the date of first documented progression or unacceptable toxicity or death.
  Interventions: Drug: FDA018-ADC
- FDA018-ADC G mg/kg (Experimental): Subjects will receive FDA018-ADC G mg/kg of body weight via intravenous (IV) infusion on Day 1 of a 14-Day cycle (Cycle 1) and on Day 1 and 8 of a 21-day cycle (Cycle 2 ~ Cycle n) in dose escalation phase, and on Day 1 and 8 of a 21-day cycle(Cycle 1 ~ Cycle n) in dose expansion phase, until the date of first documented progression or unacceptable toxicity or death.
  Interventions: Drug: FDA018-ADC

INTERVENTIONS:
Drug: FDA018-ADC — Subjects will receive an intravenous infusion of FDA018-ADC until confirmed progression, unaccepted toxicity, or any criterion for withdrawal from the study.
  Other Names: FDA018-Antibody-drug Conjugate; F0024

SUMMARY:
This is a Phase 1, open-label, dose escalation and dose expansion study to evaluate the safety, tolerability, pharmacokinetics and efficacy of FDA018-ADC in patients with advanced/metastatic solid tumors.

DETAILED DESCRIPTION:
This is a first-in-human (FIH), Phase 1, open-label, dose escalation and dose expansion study to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of FDA018-ADC in patients with advanced/metastatic solid tumors. FDA018-ADC is administered via intravenous infusion using an accelerated titration method followed by a conventional 3 + 3 study design to identify the maximum tolerated dose (MTD) and dose-limiting toxicities（DLT）during 35-day cycle with 3 doses. The expansion phase enrolled patients into three cohorts defined by tumor type: cohort 1 included patients with locally advanced or metastatic TNBC; cohort 2 included patients with non-small-cell lung cancer (NSCLC); and cohort 3 included those with other locally advanced or metastatic solid tumors. The efficacy and safety, as well as the recommended phase 2 dose (RP2D) were determined in this phase.

ELIGIBILITY:
Inclusion Criteria:

1. Patients able to give written informed consent;
2. Age ≥ 18 and ≤ 75 years old, male or female;
3. Patients have histological or cytological diagnosis with advanced solid tumors, cann't benefit from existing standard treatment options, and are not suitable for surgical resection or radiation therapy for the purpose of cure; tumor types in the study include: triple-negative breast cancer (TNBC), urothelial cancer (UC), non-small-cell lung cancer (NSCLC), small-cell lung cancer (SCLC), endometrial, gastric adenocarcinoma, esophageal, ovarian, colorectal and so on.
4. Have measurable lesions defined in RECIST v. 1.1;
5. Expected survival ≥ 12 weeks;
6. Eastern Cancer Cooperative Group (ECOG) performance status 0-1;
7. Adequate bone marrow, hepatic, and renal function;
8. All acute toxicity of previous anti-tumor treatment or surgery is relieved to baseline severity or NCI CTCAE version 5.0 ≤ 1;
9. Tumor tissue sections available；
10. Patients of child bearing potential must agree to take contraception during the study and for 6 months after the last day of treatment.

Exclusion Criteria:

1. Previous treatments for anti-Trop-2 antibody or other treatments against Trop-2, such as IMMU-132;
2. Have history of an anaphylactic reaction to irinotecan or ≥ Grade 3 GI toxicity to prior irinotecan, or previously allergic to macromolecular protein preparations;
3. Have had other malignant tumors in the past 5 years;
4. Received other anti-tumor treatments (including chemotherapy, radiotherapy, Targeted therapy, immunotherapy, experimental treatment and so on) within 4 weeks;
5. Infection requiring intravenous antibiotic use within 1 week or Fever of unknown cause occurred before the first administration> 38.5℃；
6. Have CNS (central nervous system) metastasis with clinical symptoms;
7. Any of the following cardiac criteria:

   1. Known history of severe heart disease, such as CHF≥ level 2, NYHA≥ level 2 and angina requiring medication;
   2. Clinically significant cardiac arrhythmia requiring anti-arrhythmia therapy;
   3. Hypertension not controlled by medication;
8. Have history of clinical significant active COPD, or other moderate-to-severe chronic respiratory illness present within 6 months;
9. Patients with poorly controlled diabetes;
10. Suffering from active chronic inflammatory bowel disease (ulcerative colitis, Crohn disease), and history of intestinal obstruction, or GI perforation;
11. Patients who had undergone major surgery or severe trauma within 4 weeks prior to the first dose;
12. Patients who had undergone autologous within 3 months of initiation of study treatment or allogeneic organ or stem cell transplantation within 6 months of initiation of study treatment;
13. Clinically active bacterial, fungal or viral infections (eg active hepatitis B (HBV), hepatitis C (HCV), human immunodeficiency virus (HIV), syphilis positive and so on);
14. Patients who had undergone systemic high-dose steroids within 2 weeks of initiation of study treatment;
15. Occurrence of serious venous/venous thrombosis within 1 year prior to the first dose, such as cerebrovascular accidents (including transient ischemic attack), deep vein thrombosis and pulmonary embolism;
16. Patients have history of psychotropic drug abuse, alcohol or drug abuse；
17. Women who are pregnant or lactating；
18. Any condition that is unstable or may jeopardize patient safety and its compliance with the study;
19. Other circumstances that is deemed not appropriate for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
The dose limiting toxicity ( DLT) | From first dose to the end of Cycle 1, up to 35 days.
  Evaluated according to NCI CTCAE V5.0
The maximum tolerated dose (MTD) | From first dose to the end of Cycle 1, up to 35 days.
  Maximum tolerated dose (MTD) is defined as the dose level immediately below the dose level at which 2 or more in a cohort of either 3 or 6 patients experiences a dose limiting toxicity (DLT) attributed to FDA018.
Adverse Events | From subject randomization up to 60 months
  To check the numbers of AEs happened during the course of trial.
Objective Response Rate (ORR) according to RECIST 1.1 | From subject randomization up to 60 months.
  ORR was defined as the rate an overall best response of either complete response (CR) or partial response (PR) according to RECIST1.1. CR was defined as the disappearance of all target lesions and reduction in short axis of any pathologic lymphnode to <10 mm. PR was defined as ≥ 30% decrease in the sum of diameters of target lesions, taking the baseline sum diameters.
Recommended phase II dose (RP2D) | From subject randomization up to 60 months.

SECONDARY OUTCOMES:
Time to peak (Tmax) | Up to 17 weeks.
  Tmax of Total Antibody, Total SN-38, Free SN-38, SN-38 Glucuronide and FDA018-ADC will be measured.
Half-life time (t1/2) | Up to 17 weeks.
  t1/2 of Total Antibody, Total SN-38, Free SN-38, SN-38 Glucuronide and FDA018-ADC will be measured.
Peak Plasma Concentration (Cmax) | Up to 17 weeks.
  Cmax of Total Antibody, Total SN-38, Free SN-38, SN-38 Glucuronide and FDA018-ADC will be measured.
Area under the plasma concentration versus time curve (AUC) | Up to 17 weeks.
  AUC of Total Antibody, Total SN-38, Free SN-38, SN-38 Glucuronide and FDA018-ADC will be measured.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From subject randomization up to 60 months.
  The subject's ADA positive rate will be assessed By ELISA.
Progression free survival(PFS) according to RECIST 1.1 | From subject randomization up to 60 months.
  Progression-free survival (PFS) was defined as the interval from the first dose start date to the date of disease progression defined as documented progressive disease (PD) or death from any cause, whichever occurs first.
Duration of Response(DOR) according to RECIST 1.1 | From subject randomization up to 60 months.
  Duration of Response was defined as the duration of overall response measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Overall Survival (OS) according to RECIST 1.1 | From subject randomization up to 60 months.
  Overall survival was defined as the time from the date of the first dose start date to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, Doctor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] Ponde N, Aftimos P, Piccart M. Antibody-Drug Conjugates in Breast Cancer: a Comprehensive Review. Curr Treat Options Oncol. 2019 Apr 1;20(5):37. doi: 10.1007/s11864-019-0633-6. PMID 30931493
- [Background] Zaman S, Jadid H, Denson AC, Gray JE. Targeting Trop-2 in solid tumors: future prospects. Onco Targets Ther. 2019 Mar 1;12:1781-1790. doi: 10.2147/OTT.S162447. eCollection 2019. PMID 30881031
- [Background] Goldenberg DM, Stein R, Sharkey RM. The emergence of trophoblast cell-surface antigen 2 (TROP-2) as a novel cancer target. Oncotarget. 2018 Jun 22;9(48):28989-29006. doi: 10.18632/oncotarget.25615. eCollection 2018 Jun 22. PMID 29989029